CLINICAL TRIAL: NCT04871399
Title: Complete Mesocolic Excision With Central Vascular Ligation in Comparison With Conventional Surgery for the Right Colon Cancer: An Italian Randomized Trial
Brief Title: Complete Mesocolic Excision in Comparison With Conventional Surgery for the Right Colon Cancer
Acronym: CoME-In
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Federico II University (Other); Agnelli Hospital, Italy (Other); Ospedale della Misericordia (Other); Candiolo Cancer Institute - IRCCS (Other); Maggiore Bellaria Hospital, Bologna (Other); Università degli Studi di Ferrara (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other); Ospedale Policlinico San Martino (Other); University of Rome Tor Vergata (Other); S. Andrea Hospital (Other); European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N.110/2019/U
Record Dates: First submitted 2021-04-23; First posted 2021-05-04 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-09

CONDITIONS: Colon Cancer
Keywords: colon cancer; Right colon cancer; Complete mesocolic excision; CME; Right Hemicolectomy; Right Colectomy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Right hemicolectomy (Non-CME) (Active Comparator): Patients will undergo conventional non-CME procedure.
  Interventions: Procedure: Conventional Right hemicolectomy (Non-CME)
- Right hemicolectomy with CME+CVL (Experimental): Patients will undergo Right hemicolectomy CME+CVL procedure.
  Interventions: Procedure: Right hemicolectomy with CME+CVL

INTERVENTIONS:
Procedure: Conventional Right hemicolectomy (Non-CME) — Transecting the Ileocolic Vein and Artery close to the Superior Mesenteric Vessels without clearing the superior mesenteric vein (SMV) from the adipose tissue. Transecting the Right Colic Vein and Artery and superior right colic vein (when present) peripherally. Transecting the Right branches of the Middle Colic Vein (MCV) and the Middle Colic Artery (MCA) peripherally, without clearing the main trunk of the MCV and the MCA. The Right Gastroepiploic Vein and artery are never transacted.
  Arms: Conventional Right hemicolectomy (Non-CME)
Procedure: Right hemicolectomy with CME+CVL — Separation of the visceral fascia from the parietal fascia by sharp dissection leaving intact mesocolon coverage. Transecting the supplying vessels at their origin from the main vessels, particularly:
  * The Ileocolic Vessels, The Right Colic Vessels,The superior right colic vein (when present), The Right branches of the Middle Colic Vein and of the Middle Colic Artery
  * The MCV and MCA at their origin in case of cancer of the hepatic flexure or of the proximal third of the transverse colon, as well as The Right Gastroepiploic Vessels at their origin from the gastrocolic trunk of Henle (GCTH) and the gastroduodenal artery.
  The SMV should be cleared from all adipose tissue all along its anterior surface until its intrapancreatic entrance.
  Arms: Right hemicolectomy with CME+CVL

SUMMARY:
An Italian randomized controlled trial parallel-group in patients with a malignant tumor of the right or proximal transverse colon requiring right hemicolectomy.

DETAILED DESCRIPTION:
This study aims to compare the Complete Mesocolic Excision With Central Vascular Ligation (CME+CVL) with the standard (non-CME) right hemicolectomy in patients with right or proximal transverse colon cancer stage II-IV(AJCC 8th edition) to determine the short and long term outcomes in terms of disease-free survival (DFS) as a primary endpoint, and safety, oncologic outcomes, quality of surgery and quality of life (QoL) as secondary endpoints.

Eligible patients will be randomized with a 1:1 ratio between CME + CVL vs standard non-CME right colectomy. The randomization sequence will be generated centrally by a computed algorithm and kept concealed to investigators.

The Right colectomy with CME + CVL includes the removal of the accessory lymphovascular supply at their origins by resecting the colon and mesocolon in an intact envelope of visceral peritoneum and mesenteric fascia. Despite the surgical approach and the type of procedure adopted, the operation should be strictly conducted following the general rules for colorectal oncologic resection, particularly as concerns proximal and distal margins length and lymph node retrieval.

All surgical approaches (open, laparoscopic, or robotic) will be allowed while the type of anastomosis performed and drain placement will be up to the surgeon's discretion.

Demographic, baseline, perioperative and postoperative characteristics will be analyzed as well.

The study expected to last six and a half years, of which one and a half years for recruiting 416 patients, 208 each arm, with five years of follow-up. Patients will be followed up at 1, 4, 12, 24, 36, and 60 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists(ASA) grade I-III.
* Right colon cancer (*The right-sided location of the cancer is defined as the location from the caecum up to the proximal third of the transverse colon), preoperative assessment of tumor stage T2-T4a, any N or T any N+ according to the National Comprehensive Cancer Network(NCCN) clinical practice guidelines in oncology: colon cancer version 2.2015); no distant metastasis.
* Informed consent

Exclusion Criteria:

* Age > 85 years old.
* T1, N0
* T4b, any N
* BMI > 30.
* Metastatic disease (Abdominal and chest CT scan will be mandatory to exclude distant metastasis.)
* American Society of Anesthesiologists(ASA) grade IV.
* History of cancer in recent 5 years.
* Need for Emergency surgery.
* Infectious disease requiring treatment.
* Pregnancy.
* Use of systemic steroids.
* No history of familial adenomatous polyposis, ulcerative colitis or Crohn's disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival at 3 years | 3 Years.
  The length of time after surgery without any signs or symptoms of local or distant recurrence.

SECONDARY OUTCOMES:
Safety-Operative time. | Intraoperative
  Total time from incision to skin closure expressed in minutes.
Safety-Intraoperative blood loss. | Intraoperative
  Defined by the volume drained in cm2 into aspiration systems and weight of gauzes, calculated, subtracting the weight of the dry gauzes and volume of saline solution used for irrigation.
Safety-Intraoperative blood transfusion. | Intraoperative
  Defined as the number of red blood cells, platelets, or plasma units transfused during the intraoperative time.
Safety- Intraoperative Complications. | Intraoperative
  Defined as any deviation from the ideal intraoperative course occurring during the operative time, Using the Classiﬁcation of Intraoperative Complications(CLASSIC).
Early postoperative complications. | 30 postoperative days.
  Number of patients with any deviation from the normal postoperative course grading by The Clavien-Dindo classification.
Late postoperative complications. | From the 31st postoperative days to the end of the study.
  The number of patients with any deviation from the normal postoperative course grading by The Clavien-Dindo classification.
Safety- Length of stay. | 30 Days.
  Defined as the length of an inpatient episode of care, calculated from the day of operation to the first discharge and based on the number of nights spent in the hospital.
Safety- Postoperative mortality rate. | 30 Days.
  The all-cause death rate, within 30 days after surgery in or out of the hospital.
Overall Survival at 3 years | 3 Years.
  Defined as the time from random assignment to the date of death due to any cause.
Overall Survival at 5 years. | 5 Years.
  Defined as the time from random assignment to the date of death due to any cause.
Disease-free survival. | 5 Years.
  Defined as the length of time after Surgical treatment (CME+CVL or Conventional non-CME procedure) that the patient survives without any signs or symptoms of colon cancer.
Other Oncologic outcomes. | 30 Days.
  The number of positive, negative, and total lymph nodes harvested, Quality of surgery specimen, quality of life by EORTC specific Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Degiuli, Professor, Principal Investigator — University of Turin, Department of Oncology
Locations (14):
- Italy (14):
  - Ospedale della Misericordia, Grosseto, Arezzo
  - Ospedale Città di Sesto San Giovanni, Sesto San Giovanni, Milano
  - S. Andrea Hospital, La Spezia, Spezia
  - Candiolo Cancer Institute - IRCCS, Candiolo, Torino
  - Ospedale E. Agnelli Pinerolo, Pinerolo, Torino
  - Maggiore Bellaria Hospital, Bologna, Bologna
  - Università degli Studi di Ferrara, Ferrara
  - Ospedale Policlinico San Martino, Genova
  - Azienda Ospedaliera Universitaria Policlinico "G. Martino", Messina
  - European Institute of Oncology, Milan
  - Federico II University, Napoli
  - University of Rome Tor Vergata, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - University of Turin (AOU.San Luigi Gonzaga), Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bertelsen CA. Complete mesocolic excision an assessment of feasibility and outcome. Dan Med J. 2017 Feb;64(2):B5334. PMID 28157065
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Benz S, Tannapfel A, Tam Y, Grunenwald A, Vollmer S, Stricker I. Proposal of a new classification system for complete mesocolic excison in right-sided colon cancer. Tech Coloproctol. 2019 Mar;23(3):251-257. doi: 10.1007/s10151-019-01949-4. Epub 2019 Mar 5. PMID 30838463
- [Background] Johnson PM, Porter GA, Ricciardi R, Baxter NN. Increasing negative lymph node count is independently associated with improved long-term survival in stage IIIB and IIIC colon cancer. J Clin Oncol. 2006 Aug 1;24(22):3570-5. doi: 10.1200/JCO.2006.06.8866. PMID 16877723
- [Background] Galizia G, Lieto E, De Vita F, Ferraraccio F, Zamboli A, Mabilia A, Auricchio A, Castellano P, Napolitano V, Orditura M. Is complete mesocolic excision with central vascular ligation safe and effective in the surgical treatment of right-sided colon cancers? A prospective study. Int J Colorectal Dis. 2014 Jan;29(1):89-97. doi: 10.1007/s00384-013-1766-x. Epub 2013 Aug 28. PMID 23982425
- [Background] West NP, Kobayashi H, Takahashi K, Perrakis A, Weber K, Hohenberger W, Sugihara K, Quirke P. Understanding optimal colonic cancer surgery: comparison of Japanese D3 resection and European complete mesocolic excision with central vascular ligation. J Clin Oncol. 2012 May 20;30(15):1763-9. doi: 10.1200/JCO.2011.38.3992. Epub 2012 Apr 2. PMID 22473170
- [Background] Bertelsen CA, Bols B, Ingeholm P, Jansen JE, Neuenschwander AU, Vilandt J. Can the quality of colonic surgery be improved by standardization of surgical technique with complete mesocolic excision? Colorectal Dis. 2011 Oct;13(10):1123-9. doi: 10.1111/j.1463-1318.2010.02474.x. PMID 20969719
- [Background] Kim NK, Kim YW, Han YD, Cho MS, Hur H, Min BS, Lee KY. Complete mesocolic excision and central vascular ligation for colon cancer: Principle, anatomy, surgical technique, and outcomes. Surg Oncol. 2016 Sep;25(3):252-62. doi: 10.1016/j.suronc.2016.05.009. Epub 2016 May 20. PMID 27566031
- [Derived] Degiuli M, Aguilar AHR, Solej M, Azzolina D, Marchiori G, Corcione F, Bracale U, Peltrini R, Di Nuzzo MM, Baldazzi G, Cassini D, Sica GS, Pirozzi B, Muratore A, Calabro M, Jovine E, Lombardi R, Anania G, Chiozza M, Petz W, Pizzini P, Persiani R, Biondi A, Reddavid R. A Randomized Phase III Trial of Complete Mesocolic Excision Compared with Conventional Surgery for Right Colon Cancer: Interim Analysis of a Nationwide Multicenter Study of the Italian Society of Surgical Oncology Colorectal Cancer Network (CoME-in trial). Ann Surg Oncol. 2024 Mar;31(3):1671-1680. doi: 10.1245/s10434-023-14664-0. Epub 2023 Dec 12. PMID 38087139

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT04871399/Prot_SAP_000.pdf